CLINICAL TRIAL: NCT04487717
Title: Prospective Assessment of nProfiler® 1 on Prognosis and Chemotherapy Response for Gastric Cancer
Acronym: PREDICT
Status: Active, not recruiting | Type: Observational
Sponsor: Novomics. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NM-CTP-05
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PREDICT cohort: Patients with pathologic stage II, III advanced gastric cancer
  Interventions: Device: nProfiler I Stomach Cancer Assay Kit

INTERVENTIONS:
Device: nProfiler I Stomach Cancer Assay Kit — nProfiler I Stomach Cancer Assay Kit (Novomics Co., Korea)

SUMMARY:
Prospective assessment of nProfiler® 1 predictive test on prognosis and chemotherapy response for resectable gastric cancer

DETAILED DESCRIPTION:
1. Background: According to Global Cancer Statistics of International Agency for Research on Cancer under World Health Organization, stomach cancer is the fifth most common cancer as there were over 1 million new cases in 2018 and the third leading cause of cancer death by 783,000 people are estimated to die of stomach cancer. In Korea, gastric cancer is the most frequent cancer in 13.3% of all cancer cases by the report of Korea Central Cancer Registry in 2018. Since 2010, adjuvant chemotherapy with advanced gastric cancer stage 2 and stage 3 patients following gastrectomy has become a standard treatment through clinical validation of increasing the patient's survival rate. However, even in the second and third stages of the same stomach cancer, the biological properties may be different.
2. Purpose:

   The nProfiler® 1 Stomach Cancer Assay is a molecular diagnostic test to predict the prognosis for patients with stage Ⅱ-Ⅲ advanced gastric cancer. This study will evaluate the clinical utility of nProfiler® 1 Stomach Cancer Assay by recruiting subjects from multi centers and observing the 5-year survival rates of Low risk, Intermediate risk, High risk according to gastric cancer prognostic molecular diagnostic test.
3. Study Procedure:

   * Obtaining of informed consent form
   * Review of provider's eligibility/ Sample preparation and delivery
   * Sample criteria evaluation
   * Subject enrollment
   * Gastric cancer prognostic prediction molecular diagnostic test
   * Prognostic group result report
   * 5-yr survival follow-up
   * Statistical analysis
4. Outcome Measures:

The following efficacy outcome measures will be assessed:

* Primary efficacy outcome measure

  :High risk and low risk group's 5-yr Overall Survival(OS) rate
* Secondary efficacy outcome measure

  * High risk and Low risk group's 3-yr Disease Free Survival(DFS) rate
  * Intermediate risk group's 5-yr OS and 3-yr DFS rate
  * Subgroup analysis : Adjuvant chemotherapy benefit of Low risk (5-yr OS rate, 3 yr DFS rate)

ELIGIBILITY:
Inclusion Criteria:

1. Sample providers criteria

   * Male and female adult patients aged 19 years or over
   * Patients with histologically confirmed gastric adenocarcinoma
   * Patients with histologically confirmed stage Ⅱ or Ⅲ
   * Patients who have undergone radical gastrectomy
   * Patients who have not received neoadjuvant chemotherapy and radiotherapy
   * Patients who have undergone a radical gastrectomy and who show no evidence of residual tumors as observed with the unaided eye or through a microscope
   * Patients who have signed a written consent of the study and signed a human derived research agreement (Form 34)
2. Sample criteria

   * The formalin-fixed paraffin-embedded (FFPE) tumor specimens in storage have a tumor amount of at least 20% and therefore can be tested.
   * The quantity (not less than 400ng) and quality (A260/280 of not less than 1.8) of RNA are sufficient for analysis.

Exclusion Criteria:

1. Sample providers criteria

   * Male and female patients aged less than 19 years
   * Patients with histologically not confirmed gastric adenocarcinoma
   * Patients with histologically confirmed stage Ⅰ or Ⅳ
   * Patients who have not undergone radical gastrectomy
   * Patients who have received neoadjuvant chemotherapy or radiotherapy
   * Patients with distant or peritoneal metastasis at the time of surgery or residual tumors after surgery
   * Patients who have not signed the study's written consent and human derived research agreement (Form 34)
2. Sample criteria

   * The FFPE tumor specimens in storage have a tumor amount of less than 20% and therefore cannot be tested
   * The quantity and quality of RNA are not sufficient for analysis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 19 years or older patients with stage II, III gastric adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognostic group's 5-yr Overall Survival(OS) rate | 5 years after last registered patient
  High risk and low risk group's 5-yr Overall Survival(OS) rate

SECONDARY OUTCOMES:
Prognostic group's 3-yr Disease Free Survival(DFS) rate | 3 years after last registered patient
  High risk and Low risk group's 3-yr Disease Free Survival(DFS) rate Intermediate risk group's 5-yr Os and 3-yr DFS rate
Subgroup analysis | 3, 5 years after last registered patient
  Adjuvant chemotherapy benefit of Low risk (5-yr OS rate, 3 yr DFS rate)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, MD., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- Novomics, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No